CLINICAL TRIAL: NCT03779321
Title: Effect of Food Acceptability on Appetite Hormones' Response in Normal Weight vs. Obese Male Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Ammar Olabi, Professor, American University of Beirut Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NUT.AO.20
Record Dates: First submitted 2018-12-06; First posted 2018-12-19 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Eating Behavior
Keywords: food, acceptability, appetite, hormones, ghrelin, GLP-1
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lean panelists (Other): Lean panelists or normal weight panelists with a BMI between 18.5 and 24.9 Acceptability was assessed
  Interventions: Other: Acceptability
- Obese panelists (Other): Obese panelists with a BMI between 25 and 29.9 Acceptability was assessed
  Interventions: Other: Acceptability

INTERVENTIONS:
Other: Acceptability — Food samples two formulations (low and high acceptability levels) of custard were used as experimental meals

SUMMARY:
Male subjects with specific body characteristics were recruited for the study. Subjects did an acceptability test on custard and completed a screening questionnaire. Around 30 subjects (15 with a normal BMI and 15 obese) continued the study. At each test day, fasting blood samples were withdrawn by a registered nurse under sterile conditions. This procedure was followed by ingestion of one of the two meals within a period of 10-15 minutes. Blood samples of 5 ml were collected at fasting and after ingestion of meals. At the end, subjects were given ad lib access to cheese pizza to assess energy intake after the custard preload. Blood analysis for GLP-1, ghrelin, insulin and glucose levels were performed.

DETAILED DESCRIPTION:
Male subjects were recruited for the study based on the following criteria: age between 18 and 50, body mass index normal or obese, non-smokers, non-alcoholic, and do not take medications. Subjects did an acceptability test on custard and completed a screening questionnaire. Around 30 subjects (15 with a normal BMI and 15 obese) continued the study. Subjects were randomly assigned to one of two meals. Each of the two meals was ingested after a 3-day adaptation period. The meals had similar macronutrient composition and provided energy equivalent to 30% of the subjects' resting energy expenditure. At each test day, fasting blood samples were withdrawn by a registered nurse under sterile conditions. This procedure was followed by ingestion of one of the two meals within a period of 10-15 minutes. Blood samples of 5 ml were collected at fasting and after ingestion of meals at 15, 30, 60, 120, 180 and 240 minutes. At the end, subjects were given ad lib access to cheese pizza to assess energy intake after the custard preload. Blood analysis for GLP-1, ghrelin, insulin and glucose levels were performed.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male
* Age: 18-50 years
* Body Mass Index (BMI): 18.5-24.9 kg/m2 or 30-39.9 kg/m2
* Stable body weight for at least three months before the study with the absence of any form of dieting, food restriction or other abnormal eating behaviors (to minimize the effect of weight change on ghrelin and GLP-1 statuses)
* Agreement on the acceptability levels of the two versions (high and low acceptability) of custard

Exclusion Criteria:

* Smoking
* Substance abuse such as alcohol or drugs
* Medical or psychological illness
* Previous gastrointestinal surgery
* History of weight fluctuation (weight loss of greater than 5% within the past 3 months)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Food acceptability | Through study completion, an average of 1 year
  Food acceptability on a 9 point hedonic scale
Ghrelin | Through study completion, an average of 1 year
  Ghrelin levels measured with Enzyme-linked immunosorbent assay (ELISA) kit
GLP-1 | Through study completion, an average of 1 year
  GLP-1 levels measured with Enzyme-linked immunosorbent assay (ELISA) kit
Insulin | Through study completion, an average of 1 year
  Insulin levels measured with Enzyme-linked immunosorbent assay (ELISA) kit
Glucose | Through study completion, an average of 1 year
  Glucose levels measured using VITROS ECiQ Immunodiagnostic System

SECONDARY OUTCOMES:
Appetite | Through study completion, an average of 1 year
  Appetite score on the visual analogue scale
Energy intake at the next meal | Through study completion, an average of 1 year
  Measuring quantity of cheese pizza consumed

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Helou N, Obeid OA, Olabi A. Effect of Meal Acceptability on Postprandial Appetite Scores and Hormones of Male Participants with Varied Adiposity. Obesity (Silver Spring). 2019 Oct;27(10):1627-1633. doi: 10.1002/oby.22583. Epub 2019 Aug 14. PMID 31411376